CLINICAL TRIAL: NCT00420719
Title: Multi-Center Pivotal Study of Motor-Point Stimulation for Conditioning the Diaphragm of Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Motor-Point Stimulation for Conditioning the Diaphragm of Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synapse Biomedical (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); Johns Hopkins University (Other); Stanford University (Other)
Responsible Party: Raymond Onders, MD, University Hospitals of Cleveland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-0009-0005
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig's disease; Diaphragm for Ventilatory Assist; Diaphragm Pacing
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

INTERVENTIONS:
Device: Intramuscular diaphragm electrodes — Conditioning of the diaphragm

SUMMARY:
The overall goal of this research is to delay the respiratory decline of patients with Amyotrophic Lateral Sclerosis (ALS) thereby increasing their lifespan by conditioning the diaphragm with laparoscopically placed electrodes.

This device currently holds an Investigational Device Exemption No. G040142 in the United States and is currently undergoing clinical trials at University Hospitals (Cleveland), Johns Hopkins, Mayo Clinic Jacksonville, California Pacific Medical Center (CPMC), Henry Ford Health System, The Methodist Hospital, and Stanford University.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and efficacy of the NeuRX RA/4 Diaphragm Pacing Stimulation (DPS) System in conditioning the diaphragm of an ALS patient to improve the quality of life and slow the progression to respiratory failure.

Amyotrophic Lateral Sclerosis (ALS, also known as Lou Gehrig's disease or Motor Neuron Disease) is a progressive neurodegenerative disease of unknown cause. One of the most important effects of progressive neuromuscular weakness in patients with ALS is the effect on respiration. Although ALS has no direct effect on the lung, it has devastating effects on mechanical function of the respiratory system. ALS affects all of the major respiratory muscle groups: upper airway muscles, expiratory muscles, and inspiratory muscles. Therefore, all patients with ALS are at significant risk for respiratory complications. Progressive inspiratory muscle weakness in ALS inevitably leads to carbon dioxide retention, inability to clear secretions and hypercarbic respiratory failure, the major cause of death in ALS.

Synapse Biomedical, in conjunction with Case Western Reserve University and University Hospitals of Cleveland, have evaluated activating the diaphragm with percutaneous intramuscular electrodes implanted laparoscopically. This eliminates any direct contact with the phrenic nerve, allows all circuitry and electronics to remain outside the body, and provides direct, selective activation to each hemidiaphragm. The NeuRx-RA/4 DPS System provides an electrical signal to the motor point of the muscle that causes the diaphragm to contract and allows patients to breathe more naturally.

The NeuRx RA/4 DPS System has been implanted in over 10 individuals with ALS, in a pilot study at the University Hospitals of Cleveland that began January, 2005.

The NeuRx RA/4 DPS System platform, also used for respiratory support for individuals with high-level spinal cord injury, has over 56 years of cumulative active implantation time. The longest term patient was implanted March 6, 2000 and has been using the DPS System as his sole means of respiratory support for over six years.

Given patient results to date the data supports safety and efficacy to proceed to pivotal study in this patient population. With no unexpected significant adverse events reported, the NeuRx RA/4 DPS System has performed reliably and safely.

Device Description: The NeuRx RA/4 Respiratory System is manufactured by Synapse Biomedical. The NeuRx RA/4 System comprises the following components: an external, battery powered Stimulator Device, an associated Programmer/Controller, Intramuscular Electrodes, associated percutaneous Lead Wires, a Surgical Placement Tool Set, and a surgical Mapping Station.

Inclusion Criteria:

* Age 18 or older
* Participants with familial or sporadic ALS diagnosed as laboratory-supported probable, probable, or definite according to the World Federation of Neurology El Escorial criteria will be eligible
* Bilateral phrenic nerve function clinically acceptable as demonstrated by bilateral diaphragm movement with fluoroscopic sniff test or with EMG recordings and nerve conduction times
* Forced Vital Capacity (FVC) between 50 - 85% of predicted values to begin screening procedures.
* FVC greater than 45% of predicted value at time of surgery.
* No underlying cardiac or pulmonary diseases that would increase the risk of general anesthesia greater than the expected risk of the patient with ALS
* Negative pregnancy test in females of child-bearing potential
* Informed consent from patient or designated representative

Exclusion Criteria:

* Preexisting implanted electrical device such as pacemaker or cardiac defibrillator.
* Underlying pulmonary diseases that were present prior to ALS that would effect pulmonary tests independent of ALS.
* Active cardiovascular disease that would increase the risk of general anesthesia
* Current pregnancy or breastfeeding
* Hospitalization for a treated active infection within the last 2 months
* Significant decision making incapacity preventing informed consent by the subject due to a major mental disorder such as major depression or schizophrenia, or dementia such as having Alzheimer's disease.
* Marked obesity

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Participants with familial or sporadic ALS diagnosed as laboratory-supported probable, probable, or definite according to the World Federation of Neurology El Escorial criteria will be eligible
* Bilateral phrenic nerve function clinically acceptable as demonstrated by bilateral diaphragm movement with fluoroscopic sniff test or with EMG recordings and nerve conduction times
* Forced Vital Capacity (FVC) between 50 - 85% of predicted values to begin screening procedures.
* FVC greater than 45% of predicted value at time of surgery.
* No underlying cardiac or pulmonary diseases that would increase the risk of general anesthesia greater than the expected risk of the patient with ALS
* Negative pregnancy test in females of child-bearing potential
* Informed consent from patient or designated representative

Exclusion Criteria:

* Preexisting implanted electrical device such as pacemaker or cardiac defibrillator.
* Underlying pulmonary diseases that were present prior to ALS that would effect pulmonary tests independent of ALS
* Active cardiovascular disease that would increase the risk of general anesthesia
* Current pregnancy or breastfeeding
* Hospitalization for a treated active infection within the last 2 months
* Significant decision making incapacity preventing informed consent by the subject due to a major mental disorder such as major depression or schizophrenia, or dementia such as having Alzheimer's disease.
* Marked obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The DPS System will slow the decline of pulmonary function, as defined by percent predicted forced vital capacity (FVC) to 30% of normal, by approximately 12 months | After completion of the study

SECONDARY OUTCOMES:
Adverse events from implantation and use of the DPS System will be logged and qualitatively compared to adverse event rates in similar patient populations. | After completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Onders, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (8):
- United States (7):
  - Forbes Norris - California Pacific Medical Center (CPMC), San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University Hospitals Of Cleveland, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
- Groupe Hospitalier Pitie-Salpetriere, Paris, France

REFERENCES:
- [Derived] Gonzalez-Bermejo J, Morelot-Panzini C, Salachas F, Redolfi S, Straus C, Becquemin MH, Arnulf I, Pradat PF, Bruneteau G, Ignagni AR, Diop M, Onders R, Nelson T, Menegaux F, Meininger V, Similowski T. Diaphragm pacing improves sleep in patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2012 Jan;13(1):44-54. doi: 10.3109/17482968.2011.597862. Epub 2011 Oct 24. PMID 22023158